CLINICAL TRIAL: NCT03615209
Title: Effekte Der Transkutanen Aurikularen Vagus-Nervenstimulation (tVNS) Auf Die Postprandiale Stoffwechselregulation im Menschen
Brief Title: Effect of Vagus Stimulation on Peripheral Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 608/2017BO1
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-07

CONDITIONS: Insulin Resistance; Glucose Intolerance
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transauricular vagus nerve stimulation (Active Comparator): Non invasive vagus nerve stimulation will be conducted with Cerbomed NEMOS via the left ear.
  Interventions: Device: Transauricular vagus nerve stimulation
- Transauricular sham stimulation (Sham Comparator): Non invasive sham stimulation will be conducted with Cerbomed NEMOS via the left ear lobe.
  Interventions: Device: Transauricular sham stimulation

INTERVENTIONS:
Device: Transauricular vagus nerve stimulation — Stimulation will be performed for 150 minutes (throughout the entire OGTT).
  Arms: Transauricular vagus nerve stimulation
Device: Transauricular sham stimulation — Sham stimulation will be performed for 150 minutes (throughout the entire OGTT)
  Arms: Transauricular sham stimulation

SUMMARY:
Two important mechanisms play a major role in the pathogenesis of type 2 diabetes: insulin resistance of the target tissues and the impaired insulin secretion from pancreatic β-cells. Postprandial factors (such as insulin) are perceived by the human brain and induce signals that regulate glucose metabolism via the parasympathetic nervous system.

Transcutaneous auricular vagus nerve stimulation (tVNS) can be used on the outer ear to stimulate the auricular branch of the vagus nerve in humans. Heart rate variability (HRV) in healthy people can be significantly increased via tVNS, indicating a shift from sympathetic activity to parasympathetic activity.

The hypothesis is that this postprandial shift results in a change in peripheral glucose metabolism. In turn, the increased parasympathetic activity could potentially result in a change in postprandial insulin sensitivity or secretion.

To test this hypothesis, this study investigates the effect of vagal stimulation versus sham stimulation on insulin sensitivity, on insulin secretion, glucose tolerance, resting energy expenditure, and on parasympathetic tone (analysis of heart rate variability).

ELIGIBILITY:
Inclusion Criteria:

* HbA1c <6.5%
* Must be able to understand the explanations of the study and the instructions

Exclusion Criteria:

* Any relevant (according to investigator's judgment) cardiovascular disease
* Neurological and psychiatric disorders
* Diabetes mellitus
* Active implants (e.g. pacemaker, cochlear implant, cerebral shunt)
* asthma
* skin diseases on the ear

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Whole body insulin sensitivity | 0-120 min
  Insulin sensitivity will be assessed by a 75g OGTT.

SECONDARY OUTCOMES:
Insulin secretion | 0-120 min
  Insulin secretion will be assessed by a 75g OGTT
Glucose tolerance | 0-120 min
  Glucose tolerance will be assessed by a 75g OGTT
Resting energy expenditure | 140-160 min. after start of stimulation
  Resting energy expenditure will be assessed by indirect calorimetry
Heart rate variability | -30 - 120 min
  Heart rate variability will be assessed from continuous ecg recordings

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heni, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
Due to ethical restrains, we will not be able to share patient level data.